CLINICAL TRIAL: NCT06969391
Title: Representation of Diet in the Management of Type 2 Diabetes in Migrant Patients at CHSD
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Other Study IDs: 0049_ENDOCRINOLOGIE
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Type 2 Diabetic Migrants Group

SUMMARY:
This observational and monocentric study aims to explore how migrant patients with type 2 diabetes perceive and represent food in the context of their diabetes care. Conducted at the Centre Hospitalier de Saint-Denis, the study investigates the cultural, social, and personal factors that influence dietary habits and how these perceptions affect the management of their condition. The goal is to improve the understanding of patient behaviors and support more culturally adapted care strategies.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic for at least 3 months
* Arrived in France less than 7 years ago
* Adult patient (age 18)
* Speaking French or English

Exclusion Criteria:

* Minor patient (age < 18 years)
* Type 1 diabetes
* Does not speak French or English
* Patient who has expressed opposition to the use of his data, or his refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study participants will be selected from patients diagnosed with type 2 diabetes who are attending the Centre Hospitalier St Denis. Specifically, the target population includes:
  Adults aged 18 years or older.
  Migrants who have arrived in France within the past 7 years.
  Type 2 diabetes diagnosis for at least 3 months.
  French or English language proficiency to facilitate communication during interviews.
  The population will primarily consist of migrants from socioeconomically disadvantaged backgrounds, including those who may face barriers such as language differences, cultural challenges, and limited access to healthcare. Participants will have a range of cultural backgrounds, as the study aims to explore how migration and cultural factors influence their understanding and management of type 2 diabetes, particularly in relation to food and diet.
  This population is chosen to address the knowledge gap regarding how migrant populations perceive and integrate dietary advice in the
Sampling Method: Non-Probability Sample
Enrollment: 11 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Representation of food in the care of diabetes in migrants Description | enrollment
  This measure will assess how migrants perceive and integrate food-related recommendations and dietary advice in the management of their type 2 diabetes. Through semi-structured interviews, the study will evaluate whether the food-related aspects of care are understood, accepted, and applied in practice by the migrant population, considering cultural and socio-economic factors.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier (CH) de Saint-Denis, Saint-Denis, France

IPD SHARING:
Plan to Share IPD: No